CLINICAL TRIAL: NCT04244695
Title: Efficacy of Oral Corticosteroid in Controlling Pain After Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Oral Steroid in Controlling Pain After TKA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, membership, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OrthoTU11
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Pain, Acute
Keywords: oral corticosteroid; postoperative pain; dexamethasone; total knee arthroplasty
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexamethasone 16 mg (Experimental): Dexamethasone (4mg) 4 tab oral once daily in the morning
  Interventions: Drug: Dexamethasone Oral
- Dexamethasone 8 mg (Active Comparator): Dexamethasone (4mg) 2 tab and placebo 2 tab oral once daily in the morning
  Interventions: Drug: Dexamethasone Oral
- Placebo (Placebo Comparator): Placebo 4 tab oral once daily in the morning
  Interventions: Drug: Dexamethasone Oral

INTERVENTIONS:
Drug: Dexamethasone Oral — To compare oral dexamethasone 16 mg vs 8 mg vs placebo in pateints undergoing unilateral TKA

SUMMARY:
To compare efficacy of oral steroid in controlling pain after TKA

DETAILED DESCRIPTION:
To compare pain and functional outcome for oral dexamethasone 16 mg, 8 mg and pacebo in patient undergoing unilateral primary total knee arthroplasy

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis of the knee who undergoing unilateral TKA
* ASA class I-III
* Informed consent
* Good cognitive function

Exclusion Criteria:

* Uncontrolled DM (HbA1C > 7)
* Uncontrolled HT
* Morbid obesity (BMI > 40)
* History of bleeding in GI tract
* Corticosteroid used within 6 months
* Sever liver or renal impairments
* Studied drug allergy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pain level | 12, 24 ,36, 48, 60 and 72 hours after surgery
  VAS for pain (0-100) at rest and on motion

SECONDARY OUTCOMES:
nausea and vomiting | in the first 72 hours after surgery
  rate of nausea and vomiting
Range of motion of the knee | 24, 72 hours then 2, 6, 12 weeks after surgery
  Flexion and extension angle
Functional outcome | 2, 6,12 weeks after surgery
  Modified WOMAC score
Blood sugar | At 8.00 am of 1, 2, 3 days after surgery
  Fasting blood sugar level
inflammatory level | At 8.00 am of 1, 2, 3 days and 2 weeks after surgery
  C-reactive protein level
Wound complications | 3 months after surgery
  Deep and superficial wound infection, wound dehiscense

CONTACTS AND LOCATIONS:
Locations (1):
- department of orthopaedic surgery, Faculty of medicine, Thammasat university, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No